CLINICAL TRIAL: NCT07103083
Title: A Randomized, Crossover, Controlled Trial Investigating the Effects of Different Cranberry-Based Beverages on Postprandial Glucose, Insulin, and GLP-1
Brief Title: Postprandial Response to Fruit Juice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean Spray Cranberries, Inc. (Industry)
Collaborators: Biofortis Innovation Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2508
Record Dates: First submitted 2025-07-09; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Blood Glucose; Blood Insulin
Keywords: fruit juice; blood glucose; metabolic health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- First product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Beverage 1; Dietary Supplement: Beverage 2; Dietary Supplement: Beverage 3; Dietary Supplement: Beverage 4; Dietary Supplement: Beverage 5; Dietary Supplement: Beverage 6
- Second product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Beverage 1; Dietary Supplement: Beverage 2; Dietary Supplement: Beverage 3; Dietary Supplement: Beverage 4; Dietary Supplement: Beverage 5; Dietary Supplement: Beverage 6
- Third product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Beverage 1; Dietary Supplement: Beverage 2; Dietary Supplement: Beverage 3; Dietary Supplement: Beverage 4; Dietary Supplement: Beverage 5; Dietary Supplement: Beverage 6
- Fourth product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Beverage 1; Dietary Supplement: Beverage 2; Dietary Supplement: Beverage 3; Dietary Supplement: Beverage 4; Dietary Supplement: Beverage 5; Dietary Supplement: Beverage 6
- Fifth product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Beverage 1; Dietary Supplement: Beverage 2; Dietary Supplement: Beverage 3; Dietary Supplement: Beverage 4; Dietary Supplement: Beverage 5; Dietary Supplement: Beverage 6
- Sixth product order: order not stated to protect study blinding (Experimental): Participant will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for one visit, followed by 3-7-day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Beverage 1; Dietary Supplement: Beverage 2; Dietary Supplement: Beverage 3; Dietary Supplement: Beverage 4; Dietary Supplement: Beverage 5; Dietary Supplement: Beverage 6

INTERVENTIONS:
Dietary Supplement: Beverage 1 — Fruit juice with zero sugar
Dietary Supplement: Beverage 2 — Fruit juice with low sugar - formulation 1
Dietary Supplement: Beverage 3 — Fruit juice with low sugar - formulation 2
Dietary Supplement: Beverage 4 — Fruit juice with full sugar
Dietary Supplement: Beverage 5 — Fruit juice with full sugar
Dietary Supplement: Beverage 6 — Glucose control beverage

SUMMARY:
The goal of this clinical trial is to determine postprandial responses to fruit juices.

DETAILED DESCRIPTION:
Fruit juice is commonly consumed as a part of a balanced diet because of hydration, flavor, and nutrient content . Dietary Guidelines for Americans 2020-2025 recognizes 100% fruit juice as a nutrient-dense beverage that can contribute to fruit and nutrient intake . Liquid form of juices may lead to faster absorption and hormonal responses . Measuring these acute metabolic responses can help clarify the role of fruit juice in dietary patterns and metabolic health .

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 to ≤45 years of age at Visit 1.
2. BMI ≥18.5 and <30.0 kg/m2 at Visit 1.
3. Fasting capillary glucose ≤110 mg/dL at Visit 1.
4. Willing to avoid consuming high-polyphenol containing foods for 48 hours prior to each test visit.
5. Willing to abstain from alcohol consumption for 24 hours prior to each study visit.
6. Non-user of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of Visit 1, with no plans to begin use during the study period.
7. Non-habitual users (i.e., daily or almost daily) of marijuana or hemp products, including Cannabidiol (CBD)/Tetrahydrocannabinol (THC) products, and willing to abstain from use throughout the study period (topical creams/lotions are allowed).
8. Willing to maintain habitual physical activity level throughout the duration of the study.
9. Willing to maintain habitual dietary pattern throughout the duration of the study, including stable intake of current vitamins, minerals, supplements and medications not interfering with study outcomes.
10. Score of 7 to 10 on the Vein Access Scale at Visit 1.
11. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
12. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, gastrointestinal, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Clinical Investigator.
2. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Section 9.1.1).
3. Unstable use (initiation or change in dose) within 30 days of Visit 1 of antihypertensive medications.
4. Unstable use (initiation or change in dose) within 30 days of Visit 1 of thyroid hormone replacement medications.
5. Use of medications or supplements that may influence carbohydrate metabolism within 30 days of Visit 1.
6. Extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian) at the discretion of the Clinical Investigator.
7. Weight loss or gain >4.5 kg in the 60 days prior to Visit 1.
8. Currently, or planning to be, on a weight loss regimen during the study.
9. Use of weight loss medication within 90 days of Visit 1.
10. History of gastrointestinal surgery for weight reducing purposes.
11. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
12. Known allergy or sensitivity to any ingredients or potential allergens contained in the study beverages.
13. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
14. History of any major trauma or major surgical event within 60 days of Visit 1.
15. Blood donation >450 mL within 60 days of Visit 2 or plans to donate blood or plasma during the study period.
16. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential with unstable use (initiation or change in dose) within 30 days of Visit 1) of sex hormones for contraception.
17. Recent history of (within 12 months of screening; Visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
18. Exposed to any non-registered drug product within 30 days prior to Visit 1.
19. Any condition the Clinical Investigator believes would interfere with the participant's ability to provide informed consent or comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Blood glucose iAUC - 2 hours | 2 hours
  Glucose incremental area under the curve (iAUC) from pre-product consumption to 120 min

SECONDARY OUTCOMES:
Blood glucose maximal concentration | 2 hours
  Plasma glucose maximal concentration (Cmax)
Blood glucose time to max concentration | 2 hours
  Plasma glucose time to Cmax
Blood glucose change | 2 hours
  Plasma glucose concentration change from (C-max) - (C-baseline))
Blood insulin iAUC | 2 hours
  Serum insulin incremental area under the curve (iAUC) from pre-product consumption to 120 min
Blood insulin maximal concentration | 2 hours
  Serum insulin maximal concentration (C-max)
Blood insulin time to max concentration | 2 hours
  Serum insulin time to C-max
Blood insulin change | 2 hours
  Serum insulin concentration change from (C-max - (C-baseline))
GLP-1 iAUC | 2 hours
  GLP-1 incremental area under the curve (iAUC) from pre-product consumption to 120 min
GLP-1 Maximal Concentration | 2 hours
  GLP-1 maximal concentration (C-max)
GLP-1 Time to Max Concentration | 2 hours
  GLP-1 time to C-max
GLP-1 Change | 2 hours
  GLP-1 concentration change from (C-max - (C-baseline))

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Antoo, MD, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No